CLINICAL TRIAL: NCT06845306
Title: Indocyanine Green Near-infrared Fluorescence Bowel Perfusion Quantitative Assessment to Prevent Anastomotic Leakage in Colorectal Surgery: a Multicentre, Randomised, Controlled Study
Brief Title: The Use of Indocyanine Green Near-infrared Fluorescence for Bowel Perfusion Quantitative Assessment in Order to Prevent Anastomotic Leakage in Colorectal Surgery
Acronym: ICG-NIRF
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vadim Kuznetsov (Network)
Responsible Party: Sponsor-Investigator, Vadim Kuznetsov, The doctor is a researcher, the BELOOSTROV Clinic of High Technologies
Organization: the BELOOSTROV Clinic of High Technologies (Network)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TBELOSTROVCOFHICG
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-01

CONDITIONS: Colo-rectal Cancer; Colonic Neoplasms Malignant
Keywords: ICG-guided quantitative assessment of bowel perfusion
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: multicentre randomized controlled trial
Who Masked: Participant
Masking Description: Intraoperative imaging cannot blind the surgeon. The patient is only blinded prior to surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The ICG group (Active Comparator): The ICG group, where, before creating the anastomosis, intestinal blood flow will be assessed using quantitative near-infrared fluorescence imaging using indocyanine green.
  Interventions: Drug: ICG-guided bowel perfusion assessment
- The control group (Placebo Comparator): The control group, where before the creation of the anastomosis, the intestinal blood flow will not be assessed.
  Interventions: Other: Conventional Bowel Anastomosis group

INTERVENTIONS:
Drug: ICG-guided bowel perfusion assessment — ICG will be injected before anastomosis is created, to quantitatively assess the perfusion status of the bowel.
  Arms: The ICG group
Other: Conventional Bowel Anastomosis group — conventional perfusion assessment
  Arms: The control group

SUMMARY:
Anastomotic leakage (AL) is a serious complication after surgery for colon cancer, leading to a significant increase in mortality.Intraoperative fluorescence imaging using indocyanine green has proven to be a feasible and reproducible technique for real-time perfusion assessment.

An increasing number of studies are being published on the use of indocyanine green (ICG) fluorescence imaging in colorectal cancer surgery, showing promising results.

Therefore, we propose conducting a multicenter, randomized controlled trial to investigate the potential use of quantitative assessment of near-infrared fluorescence imaging with indocyanine green (ICG) to prevent anastomotic leaks during colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years old
* ECOG status 0-2
* Written informed consent
* histologically confirmed neoplasms malignant of the colon (caecum, ascending, transverse, descending, sigmoid)
* Scheduled for colorectal resection with primary anastomosis

Exclusion Criteria:

* Pregnancy or breast feeding
* Colon obstruction, perforation or bleeding complicating the tumor
* Medical contraindications for surgical treatment
* Known allergy or history of adverse reaction to ICG, iodine or iodine dyes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1268 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
30-days Anastomotic Leakage (AL) rate | 30-days
  Anastomotic leakage rate

SECONDARY OUTCOMES:
complication rate | 30-days
mortality | 30-days
days in hospital stay | 90-days

CONTACTS AND LOCATIONS:
Overall Officials: Victor Kashchenko, Doctor of Medical Sciences, Study Director — BELOOSTROV Clinic of High Technologies
Locations (1):
- BELOOSTROV Clinic of High Technologies, Vsevolozhsk District, Leningradskaya Oblast', Russia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF